CLINICAL TRIAL: NCT04666558
Title: Heal-Me PiONEeR (Personalized Online Nutrition and Exercise Routines) - Reconnecting Vulnerable Outpatients With Multidisciplinary Care - a Randomized Controlled Trial Assessing 3 Levels of Online Programming in the Time of COVID
Brief Title: Heal-Me Personalized Online Nutrition and Exercise Routines
Acronym: PiONEeR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00103715
Record Dates: First submitted 2020-11-30; First posted 2020-12-14 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-07

CONDITIONS: Cancer; Lung Diseases; Liver Diseases
Keywords: Exercise; Nutrition; Chronic Disease; Virtual
MeSH Terms: conditions — Neoplasms; Lung Diseases; Liver Diseases; Motor Activity; Chronic Disease | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care (No Intervention): The standard of care response to COVID. Educational materials will be provided to patients via email. The package will include a combination of personalized exercises, and nutrition information for healthy eating. Participants will also receive a Garmin watch to track their activity over the intervention.
- App-Based, Personnel-Light Care (Experimental): An app-based, "personnel-light" approach to virtual care with a focus on support through group-based interactions with the Trainers, Dietitians and other participants. The patient's personalized 12-week home based exercise program will be enabled in the app after a baseline exercise specialist appointment. The 10-week nutrition program will be enabled at week 3 after a virtual dietitian assessment in week 2 (~1 hour). The home programs will auto-progress. Participants will also receive a Garmin watch to track their activity over the intervention.
  Interventions: Other: Exercise & Nutrition
- App-Based, Personnel-Intensive Care (Experimental): An app-based, "personnel-intensive" approach to virtual care with support through a combination of group-based interactions with Trainers, Dietitians and other participants, as well as one-on-one support with Exercise Trainers and Dietitians. In addition to Group 2 features, patient interaction with Trainers will be via live group classes AND 1-to-1 sessions: up to seven 1-to-1 consultations with an exercise specialist and three 1-to-1 consultations with a dietitian to review progress and goals and make any necessary modifications to programming. Participants will also receive a Garmin watch to track their activity over the intervention.
  Interventions: Other: Exercise & Nutrition

INTERVENTIONS:
Other: Exercise & Nutrition — App-based live group exercise classes, personalized follow-up asynchronous workouts, live group nutrition classes, and protein tracking.
  Arms: App-Based, Personnel-Light Care
Other: Exercise & Nutrition — App-based live group exercise classes, personalized follow-up asynchronous workouts, live group nutrition classes, and protein tracking. Additional one-one-one exercise and nutrition support is provided too.
  Arms: App-Based, Personnel-Intensive Care

SUMMARY:
The purpose of this study is to compare 12-weeks of virtual multidisciplinary programming provided at three levels of support intensity to determine impacts on clinical outcomes, acceptability, and cost amongst outpatients with cancer, liver disease, or lung disease.

Participants will be randomized to one of three groups: (i) standard care, (ii) a personnel-light app-based intervention, (iii) a personnel-intensive app-based intervention. Participants randomized to standard care will receive exercise and nutrition resources as well as a Garmin watch. Participants in the experimental groups will receive standard care, plus a 12-week multidisciplinary app-based personalized program involving 12 weeks of exercise programming and 10-weeks of nutrition programming. Participants in study group 3 will receive additional one-on-one care.

The Research Ethics Board at the University of Alberta has approved this study. The protocol will measure patient-related outcome measures including physical function, quality of life, social isolation, and anxiety, as well as measures of acceptability and cost. 216 participants will take part in this study (n=72 per arm).

Analyses: fitness testing and patient-reported outcomes will be administered before and after the intervention. Fitness and patient-reported outcomes will be compared using linear mixed models with random effects. App acceptability will be compared between groups using Chi-Square.

DETAILED DESCRIPTION:
INTRODUCTION:

COVID-19 related social distancing have a profound impact on vulnerable people living with chronic conditions, including cancer and organ failure. Pre-pandemic, many of these patients relied on and benefited from multidisciplinary supports and structured programming to maintain well-being and function. Many of these in-person supports are not currently available, which has disconnected these patients from the care they need to stay well.

Virtual modalities are a promising solution that allow multidisciplinary programs (i.e. exercise and nutrition) to continue to deliver support for these patients when social distancing doesn't allow these programs to run in-person. However, it's currently unclear whether virtual programming is acceptable in these populations, and what level of support is best in terms of benefits and costs.

The purpose of this study is to compare 12-weeks of virtual multidisciplinary programming provided at three levels of support intensity to determine impacts on clinical outcomes, acceptability, and cost amongst outpatients with cancer, liver disease, or lung disease.

OBJECTIVES:

1. As compared to control, assess the impact of a 12-week virtual exercise and nutrition program (delivered at 2 levels of support) on: physical function and mental health outcomes.
2. As compared to the modeled costs of in-person programming, assess the cost of a 12-week virtual exercise and nutrition program (delivered at 2 levels of support).
3. Assess the acceptability of the virtual exercise and nutrition programming to patients and members of the study team who deliver the intervention.

METHODS:

This is a mixed-methods, 12-week randomized controlled trial with randomization to one of three study groups with increasing virtual multidisciplinary support for outpatients. Participants will include people living with one of the following three chronic conditions: cancer, lung disease, or lung or liver disease (post-transplantation).

Group 1 - The standard of care response to COVID. Educational materials will be provided to patients via email. As needed, the package will include a combination of personalized exercises, disease-tailored tips for healthy eating and COVID precautions. Ad hoc telephone or virtual contact with patients will be at the providers' discretion.

Group 2 - An app-based, "personnel-light" approach to virtual care with a focus on support through group-based interactions with the Trainers and other participants during live group exercise and nutrition classes (~3/week). The patient's personalized 12-week home based exercise program will be enabled in the app after a baseline exercise specialist appointment and the 10-week nutrition program will be enabled at week 3 after a dietitian assessment in week 2. The home programs will auto-progress.

Group 3 - An app-based, "personnel-intensive" approach. In addition to Group 2 features, patient interaction with Trainers will be via live group classes AND 1-to-1 sessions: seven 1-to-1 consultations with an exercise specialist and three 1-to-1 consultations with a dietitian to review progress and goals and make any necessary modifications to programming.

OUTCOMES & ANALYSES:

All analyses adhere to the intention-to-treat-principle (ITT). Fitness assessments and patient-reported outcomes will be collected at baseline and 12-weeks. Primary and secondary outcomes from these data will be analyzed using linear mixed models with random effects. Adherence and app acceptability (survey) will be compared between groups using the chi-square. Costs of each level of support will be compared with the cost of in-person programming using a publicly funded provincial payer perspective and will be presented in the Net Benefit framework.

Interviews will be conducted with participants, caregivers, and program instructors to determine program acceptability and barriers and facilitators. Inductive content analysis will be used to analyze qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* In one of the following 3 disease groups:

  1. Cancer survivor who has completed treatment or is receiving maintenance therapy
  2. Patient who is currently post-transplantation from liver or lung transplantation
  3. Patient with chronic lung disease who may or may not be listed for organ transplantation
* Previous enrolment in exercise rehabilitation program (i.e. rehabilitation "graduate")
* Access to an Internet connected device with video and audio capabilities

Exclusion Criteria:

* Compassionate care
* Unsafe to participate in a virtual exercise program
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Functional Scale (LEFS) | 12 Weeks
  The difference in the pre- vs post-intervention change in LEFS score between groups (score range: 0-80, higher scores indicate higher function)

SECONDARY OUTCOMES:
Upper Extremity Functional Index (UEFI) | 12 weeks
  The difference in the pre- vs post-intervention change in UEFI score between groups (score range: 0-80, higher scores indicate higher function)
Timed Sit-to-Stand (60 & 30 seconds) | 12 Weeks
  The difference in the pre- vs post-intervention change in # of repetitions completed over the Timed Sit-to-Stand between groups
Timed One-Legged Stance | 12 Weeks
  The difference in the pre- vs post-intervention change in Timed One-Legged Stance between groups
2-Minute Step Test (2MST) | 12 Weeks
  The difference in the pre- vs post-intervention change in the # of steps completed in the 2MST between groups
Sit-and-Reach | 12 Weeks
  The difference in the pre- vs post-intervention change in the sit-and-reach distance between groups
Step Count & Activity Minutes | 12 Weeks
  The difference in the pre- vs post-intervention change in step count and activity minutes (Garmin watch) between groups
Overall Well-Being (The World Health Organization-5 [WHO-5] Well-Being Index) | 12 Weeks
  The difference in the pre- vs post-intervention change in The World Health Organization-5 (WHO-5) Well-Being Index between groups (score range: 0-25, higher scores indicate higher well-being)
Resilience (10-Item Connor Davidson Resilience Scale) | 12 Weeks
  The difference in the pre- vs post-intervention change in resilience, as measures by the 10-Item Connor Davidson Resilience Scale, between groups (score range: 0-40, higher scores indicate higher resilience)
General health-related quality of life (36-Item Short Form Survey [SF-36]) | 12 Weeks
  The difference in the pre- vs post-intervention change in health-related quality of life, as measured by the SF-36, between groups (score range: 0-100, higher scores indicate a more favorable health state)
General health-related quality of life (5-Level EQ-5D [EQ-5D-5L]) | 12 Weeks
  The difference in the pre- vs post-intervention change in health-related quality of life, as measured by the EQ-5D-5L, between groups (visual analogue score range: 0-100, higher scores indicate a more favorable health state)

OTHER OUTCOMES:
Physical activity | 12 Weeks
  The difference in the pre- vs post-intervention change in proportion of "yes" answers to the single-item physical activity questionnaire from pre- to post-intervention between groups
Sedentary Time (International Sedentary Assessment Tool - ISAT) | 12 Weeks
  The difference in the pre- vs post-intervention change in sedentary time, as self-reported on the ISAT between groups
Protein Intake | 12 Weeks
  The difference in the pre- vs post-intervention change in protein intake (grams) between groups, based on 3-day food record(s)
Calorie Intake | 12 Weeks
  The difference in the pre- vs post-intervention change in calorie intake (kilocalories) between groups, based on 3-day food record(s)
Micronutrient Intake | 12 Weeks
  The difference in the pre- vs post-intervention change in micronutrient intake (milligrams) between groups, based on 3-day food record(s)
Beliefs and outcome expectations about exercise | 12 Weeks
  The difference in the pre- vs post-intervention change in the 6-item COM-B scale between groups (score range: 0-120, higher scores indicate higher capability, opportunity, motivation)
Program acceptability (Unified Theory of Acceptance and Use of Technology - UTAUT) | 12 Weeks
  The difference in the pre- vs post-intervention change in the UTAUT scale between groups (score range: 0-92, higher scores indicate higher app acceptance and use)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tandon P, Ismond KP, Purdy G, Cruz C, Etruw E, Suderman K, Hyde A, Stickland M, Spence JC, Lien DC, Bhanji R, Prado CM, Miguel-Cruz A, Joy AA, Yaskina M, McNeely ML. Acceptability and Effectiveness of a Fully Web-Based Nutrition and Exercise Program for Individuals With Chronic Disease During COVID-19: Randomized Controlled Trial. J Med Internet Res. 2025 Mar 24;27:e57537. doi: 10.2196/57537. PMID 40126542
- [Derived] Tandon P, Purdy G, Ismond KP, Cruz C, Etruw E, Suderman K, Hyde A, Stickland M, Spence JC, Lien DC, Bhanji R, Prado CM, Cruz AM, Joy AA, Yaskina M, Round J, Harback K, Padwal R, McNeely ML. Heal-me PiONEer (personalized online nutrition and exercise): An RCT assessing 2 levels of app-based programming in individuals with chronic disease. Contemp Clin Trials. 2022 Jul;118:106791. doi: 10.1016/j.cct.2022.106791. Epub 2022 May 13. PMID 35569753
- [Derived] Cruz C, Prado CM, Punja S, Tandon P. Use of digital technologies in the nutritional management of catabolism-prone chronic diseases: A rapid review. Clin Nutr ESPEN. 2021 Dec;46:152-166. doi: 10.1016/j.clnesp.2021.10.020. Epub 2021 Nov 1. PMID 34857190